CLINICAL TRIAL: NCT06937151
Title: Arthrocentesis Versus Rocabado Exercises on Temporomandibular Disc Displacement Without Reduction
Brief Title: Comparison Between Arthrocentesis and Rocabado Exercises on Temporomandibular Disc Displacement Without Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Shawkey Mohamed, Physical Therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003932
Record Dates: First submitted 2023-12-03; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Temporomandibular Joint Disorders, Articular Disc Disorder (Reducing or Non-Reducing)
Keywords: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Study group) ROCABADO APPROACH : (Active Comparator): Group A (Study group):
  This group includes thirty-four patients with temporomandibular joint disc displacement without reduction, who will receive the Rocabado approach exercise program 6×6 AND MANIPULATION
  Interventions: Procedure: Rocabado approach exercise program 6×6 and manibulation .
- Group B (Control group) ARTHOROCENTESIS: (Active Comparator): This group includes thirty-four patients with temporomandibular joint disc displacement without reduction who will receive TMJ Arthrocentesis
  Interventions: Procedure: Arthrocentesis

INTERVENTIONS:
Procedure: Rocabado approach exercise program 6×6 and manibulation . — Rocabado's approach (Rocabado's 6 × 6 Exercises and manipulation). This program included 6 exercises to be performed 6 times a day, repeated 6 times, and three gliding exercises.
  Arms: Group A (Study group) ROCABADO APPROACH :
Procedure: Arthrocentesis — Participants in the Control Group underwent arthrocentesis of the affected temporomandibular joint. The procedure was performed as follows:
  Anesthesia: Local anesthesia was administered to the area surrounding the TMJ.
  Needle Insertion: A 20-gauge needle was inserted into the upper joint space approximately 10 mm anterior to the tragus.
  Lavage: The joint was lavaged with lactated Ringer's solution to reduce inflammation and remove debris. The joint was irrigated with lactated Ringer's solution.
  Other Names: TMJ joint washing
  Arms: Group B (Control group) ARTHOROCENTESIS:

SUMMARY:
The present study will be designed to compare the short- and medium-term results of arthrocentesis and non-surgical methods Rocabado approach in early disc displacement without reduction.

DETAILED DESCRIPTION:
This study will be designed to provide a comparison between the effect of the Rocabado approach as a conservative treatment and temporomandibular joint arthrocentesis in temporomandibular joint disc displacement without reduction.

Delimitations:

This study will be delimited in the following aspects:

1. Patients:

   The study group will be composed of sixty-eight patients with temporomandibular joint disc displacement without reduction will be enrolled in the study. Group A: It will be composed of thirty-four patients with TMJ disc displacement without reduction who are started on the Rocabado approach- 4 - 6×6 exercise program. Include therapeutic exercise, and patient education focusing on the temporomandibular joint. Repeat measurements will be performed on 1st measurement at the baseline before any intervention, 2nd measurement after 8 weeks of treatment by a physiotherapist. Group B: It will be composed of thirty-four patients with disc displacement without reduction who are started on TMJ arthrocentesis procedure with medical and nursing care.
2. Equipment and tools:

2.1-Measurement equipment: Thera bite ROM scale 8-Item Jaw Functional Limitation Scale (JFLS-8) (Valid Arabic version) visual anlogue scale 2.2-Therapeutic procedures: Rocabado's 6X6 Exercise Program and manibulation

ELIGIBILITY:
Inclusion Criteria:

* History of a sudden reduction in the mandibular opening. Unassisted mandibular opening 35 mm.
* Mandibular opening with assistance increased by ≥3 mm from
* unassisted opening, with a prior history of click, click disappearance, and a sudden decrease in opening.
* Magnetic resonance imaging (MRI) diagnosis of Disc displacement without reduction.
* Persistence of the symptoms indicated in the first item for a Maximum of 3 weeks.
* clinical diagnosis of unilateral Disc displacement without reduction of the temporomandibular joint.

Exclusion Criteria:

* History of major jaw trauma.
* Dentofacial deformity.
* Psychiatric illness.
* Chronic headache. Presence of other disorders involving the TMJ.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Thera Bite RANGE OF MOTION scale | pre treatment and eight weeks post treatment
  Will be used for measuring the Maximal interincisal opening, lateral movement will be measured.
  Measuring Maximal Interincisal Opening :
  1. Patient Positioning: The patient opens their mouth as wide as possible without discomfort.
  2. Scale Placement: The range of motion scale is positioned so that the notch rests on the edge of the lower incisor.
  3. Measurement: Rotate the scale until it contacts the upper incisor, and record the reading at the point of contact.
  Measuring Lateral Excursion Movement:
  1. Scale Alignment: Rest the range of motion scale against the lower incisors with the upper and lower teeth closed together.
  2. Arrow Alignment: Align the arrow on the scale with an interproximal space between two upper teeth.
  3. Measurement: Move the mandible laterally (side-to-side) and record the measurements on the lateral side.
8-Items Jaw Functional Limitation Scale | pre treatment and eight weeks post treatment
  Disability related to orofacial pain, which makes it a generic tool that one can use it for different types of orofacial pain conditions.
  1. Preparation: Select a quiet and distraction-free environment.
  2. Understanding the Scale: Rate each item on a scale from 0 (no limitation) to 10 (severe limitation).
  3. Completing the Questionnaire: Carefully read each question and reflect on your jaw function over the past week.
  4. Items to Rate: Assess difficulties in chewing, mouth opening, and emotional expression.
  5. Time Required: Completion typically takes less than 5 minutes.
  6. Post-Completion: Higher scores indicate greater functional limitations.
Visual analog scale | pre treatment and eight weeks post treatment
  One of the pain rating scales,
  1. Preparation: Ensure the VISUAL ANALOG SCALE line is accurately printed to scale (10 cm) with endpoints labeled:
     * 0 = No pain.
     * 10 = Worst imaginable pain.
  2. Patient Instructions: Ask the patient to mark their current pain level on the line.
  3. Score Measurement and Interpretation: Measure the distance in centimeters from the "no pain" end (0) to the patient's mark to determine the score out of 10. Higher scores indicate greater pain intensity (e.g., a mark at 6 cm corresponds to a pain level of 6/10).
  4. Recall Period: Patients report either their current pain or pain experienced within the last 24 hours, depending on assessment context.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kafer Shoukr Spechialized Hospital, Banhā, Banha
  - Kafer Shoukr Spechialized Hospital, Banhā, Qalubiah

IPD SHARING:
Plan to Share IPD: No